CLINICAL TRIAL: NCT04586855
Title: Can Ultrasound Imaging of Both Upper Airways and Diaphragm Be Used to Guide Efficacy on Non-invasive Ventilation and Cough Assist
Brief Title: Ultrasound Imaging of the Larynx and Diaphragm During NIV and Cough Assist
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: St Vincent's Hospital, Sydney (Other); Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 97615
Record Dates: First submitted 2020-07-27; First posted 2020-10-14 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2021-07

CONDITIONS: Healthy Persons
Keywords: Transnasal Fiberoptic Laryngoscopy; Diagnostic Ultrasound; Cough Assist; Noninvasive ventilation
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy persons: Noninvasive ventilation and Cough Assist
  Interventions: Diagnostic Test: Diagnostic Ultrasound; Diagnostic Test: Transnasal Fiberoptic Laryngoscopy

INTERVENTIONS:
Diagnostic Test: Diagnostic Ultrasound — To investigate if Ultrasound imaging can visualize the larynx during NIV and Cough Assist, and be as accurate as laryngoscopy
Diagnostic Test: Transnasal Fiberoptic Laryngoscopy — To investigate if Ultrasound imaging can visualize the larynx during NIV and Cough Assist, and be as accurate as laryngoscopy

SUMMARY:
The study examines if diagnostic ultrasound imaging of larynx and diaphragm can be as accurate as transnasal fiberoptic laryngoscopy in visualizing the larynx during NIV and Mechanically Assisted Cough interventions.

DETAILED DESCRIPTION:
Transnasal fiberoptic laryngoscopy (TFL) is gold standard for visualising the larynx. TFL has been used to visualize the laryngeal response patterns during non-invasive therapeutic interventions, as during Mechanically Assisted Cough in patients with Amyotrophic Lateral Sclerosis. The examinations revealed that the larynx adducted during the application of positive pressures, which restricted the airflow and reduced the efficacy of the treatment. The higher treatment pressures resulted in ineffective interventions as a result of the adducted vocal cords obstructing flow. This knowledge has changed the treatment approach for patients with possible upper airway instability by individualizing the treatment pressures and flow due to laryngeal responses.

TFL may cause slight discomfort when placing the laryngoscope. Diagnostic ultrasound is non-invasive easily applicable technique that has gained increasing popularity in diagnosing cardiopulmonary and laryngeal conditions during the recent times. The aim of the study is to investigate whether the diagnostic ultrasound of the larynx can be as accurate as TFL during Mechanically Assisted Cough and Non-Invasive Ventilation (NIV). The present study will include healthy participants. Hypothesis is that diagnostic ultrasound of larynx can provide clinical valuable information of the laryngeal response patterns during Mechanically Assisted Cough and NIV.

The aims of the study are:

* To evaluate the feasibility of diagnostic ultrasound imaging of the larynx, and to compare to the gold standard of TFL used during ongoing NIV and Mechanically Assisted Cough in healthy subjects.
* To evaluate the feasibility of ultrasound imaging if the diaphragm during ongoing NIV and Mechanically Assisted Cough in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* history of laryngospasm or pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be recruited among Healthcare Professionals and medical- and physiotherapy students
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Opening movements in larynx on transnasal fiberoptic laryngoscopy (TFL) during inspiration | Day 1
  Number of participants.
Obstructive movements in larynx on TFL during inspiration | Day 1
  Number of participants.
Closure in larynx on TFL during the compression phase of cough | Day 1
  Number of participants.
Opening movements in larynx on TFL during expiration | Day 1
  Number of participants.
Narrower movements in larynx on TFL during expiration | Day 1
  Number of participants.
Obstructive movements in larynx on TFL during expiration | Day 1
  Number of participants.
Opening movements in larynx on Anterior Ultrasound (USA) during inspiration | Day 1
  Number of participants.
Obstructive movements in larynx on USA during inspiration | Day 1
  Number of participants.
Closure in larynx on USA during the compression phase of cough | Day 1
  Number of participants.
Opening movements in larynx on USA during expiration | Day 1
  Number of participants.
Narrower movements in larynx on USA during expiration | Day 1
  Number of participants.
Obstructive movements in larynx on USA during expiration | Day 1
  Number of participants.
Opening movements in larynx on Lateral Ultrasound (USL) during inspiration | Day 1
  Number of participants.
Obstructive movements in larynx on USL during inspiration | Day 1
  Number of participants.
Closure in larynx on USL during the compression phase of cough | Day 1
  Number of participants.
Opening movements in larynx on USL during expiration | Day 1
  Number of participants.
Narrower movements in larynx on USL during expiration | Day 1
  Number of participants.
Obstructive movements in larynx on USL during expiration | Day 1
  Number of participants.
Comparison of observed movements in the larynx on transnasal fiberoptic laryngoscopy (TFL) and Anterior Ultrasound (USA) imaging. | Day 1
  The chi-square test will assess differences between examination methods.
Comparison of observed movements in the larynx on transnasal fiberoptic laryngoscopy (TFL) and Lateral Ultrasound (USL) imaging. | Day 1
  The chi-square test will assess differences between examination methods.
Comparison of observed movements in the larynx on Anterior Ultrasound (USA) and Lateral Ultrasound (USL) imaging. | Day 1
  The chi-square test will assess differences between examination methods.
Ultrasound imaging of diaphragm excursion | Day 1
  Measurements will be performed in quiet breathing, NIV and Cough Assist. Diaphragm excursions are recorded in M-mode, and will be presented in millimeters.

SECONDARY OUTCOMES:
Subjects perception of the examination with TFL - VAS scale | Day 1
  Participant's experience of the examination will be evaluated on a Visual Analog Scale (VAS) from 0-10 where higher number indicate more discomfort.
Subjects perception of the examination with Laryngeal ultrasound - VAS scale | Day 1
  Participant's experience of the examination will be evaluated on a Visual Analog Scale (VAS) from 0-10 where higher number indicate more discomfort.
Airflow registration | Day 1
  A pneumotachograph inserted in the Circuit between the facemask and the therapeutic device will register airflow during the interventions. Interruptions of the airflow will verify the possible laryngeal adductions.
Pressure registration | Day 1
  A pressure transducer inserted in the Circuit between the facemask and the therapeutic device measures the pressure and verify the settings of the NIV and Mechanically assisted Cough.

CONTACTS AND LOCATIONS:
Overall Officials: Tiina M Andersen, PhD, Principal Investigator — Haukeland University Hospital; George Ntoumenopoulos, PhD, Study Chair — St Vincent's Hospital, Sydney; Maria Vollsæter, PhD, Study Chair — Haukeland University Hospital; Anne Kristine Brekka, MSc, Study Chair — Sorlandet Hospital HF; Ola D Røksund, Professor, Study Chair — Bergen University College
Locations (1):
- Haukeland University Hospital, Bergen, Vestlandet, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fernald PS, Linden JD. The human content response in the Holtzman Inkblot Technique. J Proj Tech Pers Assess. 1966 Oct;30(5):441-6. No abstract available. PMID 5339574
- [Background] Andersen TM, Sandnes A, Fondenes O, Nilsen RM, Tysnes OB, Heimdal JH, Clemm HH, Halvorsen T, Vollsaeter M, Roksund OD. Laryngeal Responses to Mechanically Assisted Cough in Progressing Amyotrophic Lateral Sclerosis. Respir Care. 2018 May;63(5):538-549. doi: 10.4187/respcare.05924. Epub 2018 Apr 17. PMID 29666294
- [Background] Brekka AK, Ntoumenopoulos G, Roksund OD, Engeset MS, Clemm H, Halvorsen T, Vollsaeter M, Andersen T. Use of Laryngeal Ultrasound to Observe Laryngeal Movements During Noninvasive Ventilation in Healthy Volunteers. Respir Care. 2025 Mar;70(3):249-257. doi: 10.4187/respcare.12201. Epub 2024 Oct 29. PMID 39472069
- [Background] Brekka AK, Vollsaeter M, Ntoumenopoulos G, Clemm HH, Halvorsen T, Roksund OD, Andersen TM. Adjustments of non-invasive ventilation and mechanically assisted cough by combining ultrasound imaging of the larynx with transnasal fibre-optic laryngoscopy: a protocol for an experimental study. BMJ Open. 2022 May 25;12(5):e059234. doi: 10.1136/bmjopen-2021-059234. PMID 35613803